CLINICAL TRIAL: NCT06223984
Title: Evaluation of the Retrospective Clinical Results of the Combined Use of Immunoglobulin and Pulse Steroid Therapies in Severe Covid-19 Patients Followed in Intensive Care Unit
Brief Title: Combined Use of Immunoglobulin and Pulse Steroid Therapies in Severe Covid-19 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Dursun Elmas, specialist doctor, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: konya city hospital,konya
Record Dates: First submitted 2024-01-23; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Pulse Steroid and Immunoglobulins Drugs in Covid 19 Patients

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group receiving standard treatment (Active Comparator): In the group receiving standard treatment, hydroxychloroquine (400 mg/day for 5 days), low moleculer weight heparin, acetylsalicylic acid, favipiravir (3200 mg on day 1, 1200 mg on days 2-5).
  Interventions: Drug: pulse steroid and nanogam
- the group receiving IVIG and pulse steroid (Active Comparator): In the IVIG and pulse steroid group, patients received pulse steroid (250 mg/day methylprednisolone for 5 days) and intravenous immunoglobulin (400 mg/kg/day for 5 days) in addition to standard treatment. The IVIG preparations given to the patients were in 100 ml volume and 10% concentration, and the commercial name was Nanogam.
  Interventions: Drug: pulse steroid and nanogam

INTERVENTIONS:
Drug: pulse steroid and nanogam — patients received pulse steroid and ivig treatments in addition to standard treatment.

SUMMARY:
In December 2019, SARS-COV-2 was isolated from patients for the first time . It then rapidly turned into a pandemic affecting the whole world.While most Covid patients survive the disease with mild symptoms, some may develop severe organ failure and respiratory failure requiring mechanical ventilation. COVİD-19 pneumonia may progress into acute respiratory distress syndrome (ARDS). The most important reason for this has been shown in studies; is thought to be because a group of patients develop a cytokine storm-associated hyperinflammatory state characterized by features of macrophage activation syndrome (MAS). The aim of this study was to evaluate the clinical outcomes of the combined use of pulse steroid and intravenous immunoglobulin therapy in patients with severe COVID-19 with severe respiratory distress in intensive care unit.

DETAILED DESCRIPTION:
In December 2019, SARS-COV-2 was isolated from patients for the first time . It then rapidly turned into a pandemic affecting the whole world.While most Covid patients survive the disease with mild symptoms, some may develop severe organ failure and respiratory failure requiring mechanical ventilation . COVİD-19 pneumonia may progress into acute respiratory distress syndrome (ARDS) , diffuse alveolar damage, and vascular endothelitis, which is comlicated with trombosis and hemorrhage. .

The most important reason for this has been shown in studies; is thought to be because a group of patients develop a cytokine storm-associated hyperinflammatory state characterized by features of macrophage activation syndrome (MAS), such as lymphopenia, elevated ferritin and elevated d-dimer. Increased proinflammatory cytokine release, especially as a result of stimulation of the immune system, has been shown to be associated with this hyperinflammatory phase .

The immune system triggered by viral infections is essential for fighting pathogens. However, the excessive production of pro-inflammatory cytokines caused by SARS-COV-2 can cause tissue damage that can lead to fatal acute respiratory distress .

Therefore, aiming to suppress the cytokine storm seems to be of critical importance for COVID-19 and similar respiratory infections that cause acute respiratory distress . Many agents have been used for this purpose, but there is no clear evidence for the management and treatment of cytokine storm.

Immunosuppression plays an important role in the treatment of cytokine storm. Studies have reported positive results of steroids used for this purpose in elderly COVID-19 patients . Various immunomodulatory agents have also been used for this purpose. In addition to treatments targeting a specific molecule such as IL-6, IL-1, agents that affect various branches of the immune inflammatory system such as intravenous immunoglobulin can be used .

The aim of this study was to evaluate the clinical outcomes of the combined use of pulse steroid and intravenous immunoglobulin therapy in patients with severe COVID-19 with severe respiratory distress in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with 2019-ncov infection confirmed by PCR;
* Absolute value of lymphocytes < 0. 6x 109/L;
* Brescia-COVID respiratory severity scale (BCRSS) score ≥3
* Hyperinflammation (defined as elevation of C-reactive protein (CRP) ≥50 mg/L or ferritin ≥500 ng/ ml)
* Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 300 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

* Age < 18
* Pregnant
* Allergic to experimental drugs
* The underlying disease is very serious and the expected survival time is less than 6 months (such as advanced malignant tumor);
* COPD or end-stage lung disease requires home oxygen therapy
* Expected survival time not exceeding 48 hours
* Autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years and older (Adult, Older Adult )
Enrollment: 178 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
absolute lymphocyte , white blood cell , neutrophil , ferritin , dimer , crp counts | on the first day of hospitalization, in the middle and at discharge from intensive care
  counts on the first day of hospitalization, in the middle and at discharge from intensive care
SOFA score | Day 1
  SOFA score at Day 1, with scores range from 0 to 24 and higher score means worse outcome
all cause mortality rate | 28 days
  died at day 28
ventilation free days | 28 days
ICU free days | 28 days
invasive and non-invasive respiratory support | 28 days
  intubated
vasopressor support | 28 days
  vasopressor support needs
renal replacement therapy | 28 days
  renal replacement therapy needs

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided